CLINICAL TRIAL: NCT01281436
Title: Health Information Technology to Support Clinical Decision Making in Obesity Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arizona State University (Other)
Collaborators: University of New Mexico (Other); University of Colorado, Denver (Other)
Responsible Party: Bonnie Gance-Cleveland, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AHRQ
Record Dates: First submitted 2011-01-14; First posted 2011-01-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Childhood Overweight; Childhood Obesity
Keywords: childhood; overweight; obesity; Health information technology; HeartSmartKids; Motivational Interviewing
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Web-based Provider training (Other): The training will include information about implementing the recommendations of the AMA, the pediatric metabolic working group, and the HEATSM guidelines into their practice setting through the use of the chronic care model for childhood obesity. Training will include self-management support, decision support, delivery-system redesign, clinical information systems, practice self-assessment, and staff development on obtaining, assessing, documenting BMI and BP; counseling families on appropriate interventions; and quality improvement processes to evaluate the practice's performance strategies.
  Interventions: Other: Web-based Provider Training
- HeartSmartKids with web-based training (Active Comparator): The providers assigned to Group 2 will receive the web-based training described in the other arm, plus the HeartSmartKids™ (HSK) system. HSK is a bilingual, HIT kiosk system with clinical decision support and tailored patient education.
  Interventions: Other: HeartSmartKids & Web-based Provider Training; Other: Web-based Provider Training

INTERVENTIONS:
Other: HeartSmartKids & Web-based Provider Training — The providers assigned to Group 2 will receive the web-based training described in the web-based training arm, plus the HeartSmartKids™ (HSK) system. HSK is a bilingual, HIT kiosk system with clinical decision support and tailored patient education.
  Arms: HeartSmartKids with web-based training
Other: Web-based Provider Training — The training will include information about implementing the recommendations of the AMA, the pediatric metabolic working group, and the HEATSM guidelines into their practice setting through the use of the chronic care model for childhood obesity. Training will include self-management support, decision support, delivery-system redesign, clinical information systems, practice self-assessment, and staff development on obtaining, assessing, documenting BMI and BP; counseling families on appropriate interventions; and quality improvement processes to evaluate the practice's performance strategies.

SUMMARY:
The purpose of this study is to address priority Research Area 3 in PAR-08-270: Health information technology (HIT) to improve health care decision making through the use of integrated data and knowledge management. The proposed study will evaluate the use of HIT for clinician decision support and tailored patient education on the implementation of the current guidelines for the prevention of obesity-related chronic conditions in health disparity populations of poor, minority youth who access care through SBHCs. The specific aims are:

1. To evaluate the effectiveness of web-based training with and without computerized clinical decision support on provider's process and outcome behaviors related to implementing the current guidelines for prevention of obesity and related conditions.

   a. Process variables include the following: i. Provider knowledge, attitudes, and barriers to implementing the guidelines. ii. Parent perception of the interpersonal process of care (i.e., provider communication, collaborative decision making, and interpersonal style).

   iii. Parent perception of provider support for their child's healthy eating and exercise.

   b. Behavior outcomes include the following: i. Provider self-reported behaviors of identification and assessment of overweight, counseling on nutrition and physical activity, use of behavioral interventions, referrals, and cultural competency.

   ii. Documentation by chart review of body mass index (BMI) percentile for age and sex; appropriate diagnosis when BMI > 85th percentile; blood pressure (BP) percentile for age, height, and sex; and ordering appropriate laboratory tests when indicated.
2. To explore the role of HIT in the processes of system change for implementation of the guidelines for prevention of obesity and related conditions, including the facilitators, barriers, and impact of the care model on change.

DETAILED DESCRIPTION:
The prevalence of overweight youth nearly quadrupled in the past four decades. An alarming increase in the number of poor, underserved, overweight minority youth is reported. This dramatic increase in overweight youth has led to the emergence of associated co-morbidities such as dyslipidemia, hypertension, type 2 diabetes, musculoskeletal disorders, respiratory conditions, and emotional problems in youth as well as increased risks of cardiovascular disease and cancer as adults. School-based health centers (SBHCs) provide access to primary care for many underserved and minority youth at risk for obesity and related chronic conditions. Primary care providers (PCPs), however, including those at SBHCs, face a number of barriers to addressing weight management in children. The rising prevalence of obesity and difficulty in identifying, assessing, and maintaining healthy weight in children and adolescents led national groups to convene expert panels that have published evidence-based guidelines. These guidelines include screening for cardiovascular risk factors and using a family-centered and culturally sensitive approach to care. The recommendations incorporate the use of motivational interviewing (MI) and the chronic care model to collaborate with families on a plan of care to improve children's health outcomes. The publication of recommendations or guidelines, however, traditionally has not changed provider behavior. Studies have shown widespread failure to follow established guidelines for a variety of conditions. The barriers to implementing guidelines include inadequate tools or resources, insufficient knowledge and skills, lack of self-efficacy, lack of time, and insufficient reimbursement. Health information technology (HIT) serves as a mechanism for providing decision support and tailored patient education materials to improve evidence-based care for the prevention of obesity and related conditions. Self-efficacy regarding obesity counseling has been linked to access to HIT. Other studies indicate that patients who received written health information with graphics that depicted their response to therapy improved their motivation to adhere to the treatment plan and were more satisfied with care. The proposed study is a comparative-effectiveness trial evaluating the impact of web-based provider training with and without HIT for provider decision support and tailored patient education. The goal is to translate into practice the current evidence-based guidelines for the prevention of obesity-related chronic conditions. HeartSmartKids™ is a decision-making tool that integrates patient health information with evidence-based guidelines and generates graphic trends of cardiovascular risks and tailored recommendations to improve patient outcomes. Elimination of health disparities in the chronic conditions related to childhood obesity depends upon the translation of best evidence into practice by the providers who care to youth at-risk for these obesity-related conditions. The unique features of this study are the SBHC setting; comparative effectiveness of web-based training on current evidence-based recommendations with and without HIT to support providers' decision making and tailored patient education; and the use of the Health Disparities Collaborative, the Institute for Healthcare Improvement's Breakthrough Series quality improvement process, and the chronic care model for childhood obesity for training providers on the current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* School Based Health Centers who serve children 5-12 years
* sees a minimum of 20 children per month for well-child care or sports physicals
* has internet access and printer
* has space for a small computer in the waiting room or check-in area
* has a primary care provider who reads English.

Inclusion criteria for parents:

* read English or Spanish

Exclusion Criteria:

* centers that have implemented the HeartSmartKids program.
* children seen for immunizations, dental, or mental health care without a well-child visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-07 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
International Life Science Institute(ILSI)Research Foundation Assessment of Overweight in Children and Adolescents | every 9-12 months
  The 35-item survey asks providers to rate themselves using a Likert-type scale on the following: (a) definitions of overweight in various age groups, (b) calculation and documentation of BMI percentile, (c) routine counseling on nutrition, physical activity, and screen time, (d) assessment of overweight children, and (e) resources and barriers that providers encounter in dealing with childhood overweight.
Chronic Care Model Elements Survey (CCMES) | every 9-12 months
  A 9-item survey that assesses the extent to which elements of the chronic care model are used in the routine care of patients in a practice. It was originally designed for patients with diabetes and was adapted for use in overweight/obesity. The total score is created as the mean of the 9 items, with the higher indicative of greater use of the elements of the CCM.

SECONDARY OUTCOMES:
Interpersonal Process of Care (IPC) | every 9-12 months
  A 29-item survey available in English and Spanish. It is a 5-point Likert-type scale that measures the patient-clinician relationship, quality, and satisfaction with care on three domains: communication, decision making, and interpersonal style. Health disparities may be attributable to differences between minorities and their counterparts in the interpersonal processes between the patients and clinicians.
Health-Care Climate Questionnaire (HCCQ) | every 9-12 months
  A measure with 6 items for eating and 6 items for regular exercise that assesses the degree of support from healthcare providers for healthy behaviors. The HCCQ for diet and exercise are scored by combining the items on each scale.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie M Gance-Cleveland, Ph.D., Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States